CLINICAL TRIAL: NCT06645951
Title: Creation, Management and Analysis of a National Database of Patients with Parathyroid Carcinoma or Atypical Parathyroid Adenoma
Brief Title: Institution of an Italian Multicenter Database of Patients with Parathyroid Carcinoma or Atypical Parathyroid Adenoma
Status: Recruiting | Type: Observational
Sponsor: F.I.R.M.O. - Fondazione Italiana Ricerca sulle Malattie dell'Osso - Ente del Terzo Settore (Other)
Responsible Party: Sponsor
Other Study IDs: 23354_oss
Record Dates: First submitted 2024-10-07; First posted 2024-10-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-10

CONDITIONS: Parathyroid Gland Carcinoma; Parathyroid Gland Atypical Adenoma
Keywords: Parathyroid carcinoma; Atypical parathyroid adenoma; Retro-prospective clinical data collection; Database of patients
MeSH Terms: conditions — Parathyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with parathyroid carcinoma: Male and female patients of any age who developed parathyroid carcinoma. The study does not include any type of intervention
- Patients with atypical parathyroid adenoma: Male and female patients of any age who developed atypical parathyroid adenoma The study does not include any type of intervention

SUMMARY:
The goal of this observational study is to create, manage and analyze a multicenter national database of patients with parathyroid carcinoma or atypical parathyroid adenoma, aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, histological, and therapeutic data in a relatively wide number of patients in Italy.

The study will include 33 specialist clinical centers of endocrinology and endocrine surgery, located throughout the Italian territory, and to which patients refer from all the 20 regions of Italy.

Data will be collected over time, both in retrospective and prospective manners, during the 10-year duration of the study, starting from the recruiting visit (basal visit) and then during each follow-up visits patients will undergo for the control of disease progression at the recruiting clinical centers.

Collected data will include both the most classic traits of the pathology and the less common ones, with the final goal of refining and deepening medical knowledge in the field of these two extremely rare parathyroid cancers and be able to define optimal clinical and therapeutic management of patients, improving their quality and life expectancy.

The main aspects this observational study aims to assess and clarify are:

1. Evaluation of prevalence and incidence of parathyroid carcinoma and atypical parathyroid adenoma in Italy, both as sporadic disease or in the context of genetic disorders.
2. Clinical, histological, and biochemical characterization of parathyroid carcinoma vs atypical parathyroid adenoma, to assess features and aspects that distinguish these two kinds of tumors and may help in the differential diagnosis.
3. Evaluation of short-term and long-term response to therapies in patients with parathyroid carcinoma and in patients with atypical parathyroid adenoma to assess possible differences between these two types of cancer and, thus, to design tailored clinical and therapeutic managements for patients.
4. Evaluation of short-term and long-term response to therapies in sporadic forms vs genetic forms of parathyroid carcinoma and atypical parathyroid adenoma, to assess possible differences between these two different forms of diseases and, thus, to design tailored clinical and therapeutic managements for patients.

The study will include two independent cohorts of female and male patients of any age, one including patients who developed parathyroid carcinoma (cohort 1) and one including patients who developed atypical parathyroid adenoma (cohort 2), both as sporadic cancer or in the context of genetic diseases. The study does not include either any control group/comparison group or healthy volunteers.

The study itself does not involve any medical intervention or drug administration. Treatments (surgery and/or drugs), for which data on response to therapy will be collected in the database, are those that are conventionally used in patients with parathyroid carcinoma or atypical parathyroid adenoma for treatment of their pathology, regardless of their inclusion in this observational study.

DETAILED DESCRIPTION:
A. Background and rationale:

Parathyroid carcinoma (PC) and atypical parathyroid adenoma (aPA) are two extremely rare forms of cancer of the parathyroid glands, that represent approximately 1% of all parathyroid tumors.

The extreme rarity of these two types of tumor results in a lack of specific and detailed clinical information on them. This, together with the current scarcity and incompleteness of multicenter and prospective studies on large case series, has not yet allowed to reach a shared consensus for the clinical and therapeutic management and follow-up of these tumors, nor the creation of specific guidelines. For this reason, the institution and management of national multicenter databases of patients with parathyroid carcinoma or atypical parathyroid adenoma are extremely important to allow the collection of a relatively high number of patients with these two endocrine cancers, whose clinical features could be, then, carefully studied in every aspect of the disease, from the most classic traits of the pathology to the less common ones, in both retrospective and prospective manners.

B. Main aim and specific objectives:

Main goal of this observational study is to create, manage and analyze a retro-prospective multicenter national database of patients with parathyroid carcinoma or atypical parathyroid adenoma in Italy, aimed at collecting and studying anamnestic, diagnostic, genetic, clinical, histological, and therapeutic data on these two extremely rare parathyroid cancers in a relatively wide number of patients.

Such a database will allow for an epidemiological evaluation of the prevalence and incidence of parathyroid carcinoma and atypical parathyroid adenoma in Italy, and to collect case history of patients whose clinical cases will be studied in detail and followed over time up to 10 years after the recruitment in the study, also as post-operative follow-up, in order to refine knowledge in the field of these two rare and malignant parathyroid tumors, to identify the most effective therapy, and direct future research in the identification of possible specific therapeutic targets.

Specific objectives of the studies are:

1. Creation of an Italian centralized multicenter database of patients with parathyroid carcinoma or atypical parathyroid adenoma, through the collection of patients at 33 specialist clinical centers of endocrinology and endocrine surgery, located throughout the Italian territory and visiting patients from all the 20 regions of Italy.
2. Collection of a relatively high number of patients with parathyroid carcinoma or atypical parathyroid adenoma, both as sporadic tumors or in the context of genetic disorders.
3. Retrospective collection of data about past clinical history of parathyroid carcinoma and atypical parathyroid adenoma, at the time of the recruiting visit.
4. Continuous and updated prospective collection of patients' data over time, starting from the first recruiting visit up to 10 years after the recruitment in the study.
5. Evaluation of the prevalence and incidence of parathyroid carcinoma and atypical parathyroid adenoma in Italy, both as sporadic disease or in the context of genetic disorders.
6. Clinical, histological and biochemical characterization of parathyroid carcinoma vs atypical parathyroid adenoma, to assess features and aspects that distinguish these two kinds of tumors and may help in the differential diagnosis.
7. Evaluation of short-term and long-term response to therapies in patients with parathyroid carcinoma and in patients with atypical parathyroid adenoma to assess possible differences between these two types of cancer and, thus, to design tailored clinical and therapeutic managements for patients.
8. Evaluation of short-term and long-term response to therapies in sporadic forms vs genetic forms of parathyroid carcinoma and atypical parathyroid adenoma, to assess possible differences between these two different forms of diseases and, thus, to design tailored clinical and therapeutic managements for patients.

C. Study population:

The study will include two independent cohorts of female and male patients of any age, one including patients who developed parathyroid carcinoma (cohort 1) and one including patients who developed atypical parathyroid adenoma (cohort 2), both as sporadic cancer or in the context of genetic diseases.

The study does not include either any control group/comparison group or healthy volunteers.

Given the extreme rarity of parathyroid carcinoma and atypical parathyroid adenoma, we estimate that we will be able to include in the study a minimum of 100 and a maximum of 300 patients affected by parathyroid carcinoma or atypical parathyroid adenoma during the 10 years of the study.

Inclusion criteria

* Cohort 1: parathyroid carcinoma
* Cohort 2: atypical parathyroid adenoma Exclusion criteria
* None

D. Study design and setting:

Non-profit, multicenter, national, retro-prospective, observational study, consisting in the design, creation, management and analysis of an Italian database of patients with parathyroid carcinoma or atypical parathyroid adenoma.

The study will last 10 years. The enrollment of patients with parathyroid carcinoma or atypical parathyroid adenoma, the inclusion in the database with retrospective collection of their clinical data, and the subsequent prospective collection of clinical follow-up data will take place throughout the duration of the study. For the retrospective collection, retrospective data on parathyroid carcinoma or atypical parathyroid adenoma will be retrieved from patient's medical records, at the time of the medical visit that the patient will carry out at the Clinical Center for the evaluation of his/her parathyroid disease, regardless of inclusion in this study. Prospective data relating to the tumor follow-up will be collected during the subsequent medical follow-up visits, scheduled for each patient as part of the clinical management of his/her parathyroid disease, regardless of inclusion in this study.

Being an observational study, this study itself does not involve the administration of any drug, nor the use of any medical device, nor does it involve additional medical visits, clinical analyses or care procedures in addition to those conventionally scheduled for the clinical and therapeutic management of patient affected by parathyroid carcinoma or atypical parathyroid adenoma. No participant biospecimens of any type will be collected and retained to perform this study. Pharmacological treatments and parathyroid surgery, for which data on response to therapy and peri-operative and post-operative outcomes will be collected in the database during the study, are those that are conventionally administered and performed in patients with parathyroid carcinoma or atypical parathyroid adenoma in the context of treatment of their pathology, regardless of their inclusion in this observational study.

All data will be collected anonymously, and they will be analyzed as aggregates. Data collected in the database will be, first, processed using descriptive statistics, such as frequency tables for categorical data, median and quartiles for quantitative data on ordinal scales and mean and standard deviation for quantitative data on metric scales. Secondly, the correlations between variables will be evaluated using the Pearson correlation index in the case of continuous variables and the chi-square test for categorical variables.

E. Data and variables:

Data collected in the database will include (if available in patient's medical records):

* Demographics (sex, year of birth)
* Family history of parathyroid carcinoma/atypical parathyroid adenoma or other parathyroid diseases in first-degree relatives
* Lifestyle habits (i.e smoke, alcohol intake)
* History of neck irradiation
* Clinical history and therapy of hyperparathyroidism prior to diagnosis of parathyroid carcinoma/atypical parathyroid adenoma
* Presence of comorbidities
* Age at diagnosis of parathyroid carcinoma/atypical parathyroid adenoma, type of diagnosis, genetic test (if performed)
* Clinical manifestations of parathyroid carcinoma/atypical parathyroid adenoma (i.e hypercalcemia, nephrolithiasis, nephrocalcinosis, bone mass loss, fragility fracture, bone pain, radiological findings of skeletal complaints, gastrointestinal manifestations)
* Pre-operative instrumental screening of the neck (neck ultrasounds, parathyroid scintigraphy with 99mTc-Sestamibi, neck CT scan, 11C-choline PET/CT, 11C-methionin PET/CT, 18F-FDG-PET/CT)
* Pre-operative biochemical measurements of parameters of parathyroid function and of bone and mineral metabolism
* Pre-operative DXA evaluation of bone status
* Pre-operative identification of lymph node and/or distant metastases
* Pharmacological therapies
* Surgical intervention (age, type, clear margins, removed lymph nodes, complications, perioperative mortality, etc)
* Post-operative histological analysis of resected tumor (surrounding tissue and vascular invasion, Ki67 index, mitotic activity, nuclear atypia, aneuploidy, immunostaining of parafibromin and other specific proteins)
* TMN tumor staging
* Somatic genetic screening of resected tumor
* Post-operative clinical follow-up (serum calcium normalization, post-operative hypoparathyroidism, episodes of hypocalcemia, episodes of hypophosphatemia, hungry bone syndrome, disease persistence, tumor recurrence, etc)
* Post-operative biochemical measurements of parameters of parathyroid function and of bone and mineral metabolism (the first check-up after parathyroid surgery, and subsequent follow-up measurements)
* Post-operative instrumental screening of the neck (neck ultrasounds, parathyroid scintigraphy with 99mTc-Sestamibi, neck CT scan, 11C-choline PET/CT, 11C-methionin PET/CT, 18F-FDG-PET/CT)
* Post-operative DXA evaluation of bone status
* Death as a consequence of carcinoma/atypical parathyroid adenoma (age of death, cause)

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: parathyroid carcinoma
* Cohort 2: atypical parathyroid adenoma

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients of any age who developed parathyroid carcinoma (cohort 1) or atypical parathyroid adenoma (cohort 2), both as sporadic disease or in the context of a genetic disorder
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2034-11-04 (Estimated); Study Completion 2034-11-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence and incidence evaluation | Through study completion, an average of 10 years
  Evaluation of prevalence and incidence of parathyroid carcinoma and of atypical parathyroid adenoma in Italy
Comparative characterization of parathyroid carcinoma and atypical parathyroid | Through study completion, an average of 10 years
  Comparative analysis of clinical, histological, and biochemical features in parathyroid carcinoma vs atypical parathyroid adenoma
Therapy response in parathyroid carcinoma and atypical parathyroid | Through study completion, an average of 10 years
  Analysis of short-term and long-term responses to treatments (surgery and/or pharmacological therapies) in parathyroid carcinoma and atypical parathyroid adenoma
Therapy response in sporadic and genetic forms of disease | Through study completion, an average of 10 years
  Analysis of short-term and long-term responses to treatments (surgery and/or pharmacological therapies) in sporadic vs genetic forms of parathyroid carcinoma and atypical parathyroid adenoma

CONTACTS AND LOCATIONS:
Locations (33):
- Italy (33):
  - U.O.C. Endocrinologia, Azienda Ospedaliero Universitaria Policlinico Consorziale, Università degli Studi di Bari "Aldo Moro", Bari
  - UOC Endocrinologia e Prevenzione e Cura del Diabete, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Dipartimento di Scienze Mediche e Chirurgiche (DIMEC), Alma Mater Studiorum Università di Bologna, Bologna
  - Endocrinologia e Diabetologia, Azienda Ospedaliero-Universitaria di Cagliari, Presidio Ospedaliero Policlinico di Monserrato, Cagliari
  - UO Endocrinologia e Malattie del Ricambio, Azienda Ospedaliero Universitaria di Ferrara, Sezione di Endocrinologia, Geriatria e Medicina Interna, Dipartimento di Scienze Mediche, Università degli Studi di Ferrara, Ferrara
  - SOD Malattie del Metabolismo Minerale ed Osseo, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Unità di Chirurgia Endocrina, Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Casa Sollievo della Sofferenza, Foggia
  - Clinica Endocrinologica, Dipartimento di Medicina Interna e Specialità Mediche (DiMI), IRCCS Ospedale Policlinico San Martino, Università di Genova, Genova
  - Clinica Pediatrica ed Endocrinologia, IRCCS Ospedale Pediatrico Giannina Gaslini, Genova
  - U.O.S.D. Centro Malattie Rare · Dipartimento di Pediatria IRCCS Ospedale Pediatrico Giannina Gaslini, Genova
  - UOC di Endocrinologia, AOU Policlinico G. Martino, Dipartimento di Patologia Umana DETEV, Università di Messin, Messina
  - Dipartimento di Malattie Endocrino-Metaboliche, IRCCS Istituto Auxologico Italiano, Milan
  - Endocrinologia Infantile, UOU di Pediatria, IRCCS Ospedale San Raffaele, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - SC Endocrinologia, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Dipartimento di Medicina Clinica e Chirurgia; Unità di Endocrinologia, Diabetologia e Andrologia; Università degli Studi di Napoli Federico II, Napoli
  - UOC di Endocrinologia e Malattie del Metabolismo, AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - SCDU Endocrinologia Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Endocrinologia, Clinica Polispecialistica San Carlo, Paderno Dugnano
  - Unità di Chirurgia Endocrina, Dipartimento di Chirurgia, Oncologia e Gastroenterologia, Università di Padova, Padua
  - UOC Endocrinologia, DIMED, Azienda Ospedaliero-Universitaria di Padova, Padua
  - Unità Operativa Endocrinologia 2, Azienda Ospedaliera Universitaria Pisana, Pisa
  - Dipartimento di Medicina Sperimentale, "Sapienza" Università di Roma, Roma - UOC Endocrinologia, Policlinico Umberto I di Roma, Roma
  - Unità di Endocrinologia e Andrologia, Dipartimento di Medicina Clinica e Molecolare, AOU Sant'Andrea, Centro di eccellenza ENETS, Università Sapienza di Roma, Roma
  - UOC Patologie osteo-metaboliche e della tiroide, Fondazione Policlinico universitario Campus Bio-Medico, Roma
  - UOC di Endocrinologia, Diabetologia e Andrologia Medica, IRCCS Humanitas Research Hospital, Rozzano
  - Donatello Bone Clinic, Casa di Cura Villa Donatello, Sesto Fiorentino
  - Dipartimento di Scienze Mediche, Chirurgiche e Neuroscienze, Policlinico Santa Maria delle Scotte, Università di Siena, Siena
  - SCDU Endocrinologia Diabetologia e Malattie del Metabolismo, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - SCDU Endocrinologia Oncologica, AOU Città della Salute e della Scienza di Torino, Università di Torino, Torino
  - IRCCS Materno-Infantile Burlo Garofolo, Trieste
  - SOC Endocrinologia, Azienda Sanitaria-Universitaria Friuli Centrale, Udine
  - UOS di Endocrinologia, Policlinico GB Rossi, Azienda Ospedaliera Universitaria Integrata di Verona, Verona